CLINICAL TRIAL: NCT00122096
Title: Preoperative Valdecoxib: CNS Penetration and Effects on Biochemical Markers of Pain and Sensitization
Brief Title: Perioperative Inflammation and Cyclooxygenase 2 (COX-2)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDK001
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Neurosurgery; Pain
Keywords: neurosurgery; COX-2; inflammation; pain
MeSH Terms: conditions — Pain; Inflammation | interventions — valdecoxib

INTERVENTIONS:
Drug: valdecoxib

SUMMARY:
Surgery initiates a complex cascade of events involving the release of chemical compounds from nerve endings and damaged tissue which leads to an inflammatory and pain response. The purpose of this investigation is to measure various chemical mediators in the blood and cerebrospinal fluid, and to test the hypothesis that they will be decreased in patients treated with a COX-2 inhibitor.

DETAILED DESCRIPTION:
Surgery initiates a complex cascade of events involving the release of nociceptive compounds from nerve endings and damaged tissue which leads to an inflammatory and hyperalgesic response. COX-2 inhibitors are often used for treating pain. This is a double-blind randomized study in surgical patients receiving a spinal drain for surgical purposes. The hypothesis is that valdecoxib will reach therapeutic concentrations in CSF, and will decrease plasma and CSF concentrations of inflammatory mediators. Subjects will receive valdecoxib 40 mg or placebo approximately 1 hr prior to surgery. Serial blood and CSF samples will be obtained. Valdecoxib and cytokine concentrations will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery requiring lumbar drain placement

Exclusion Criteria:

* Contraindication to COX-2 inhibitor (renal or hepatic insufficiency)
* Known adverse reaction to nonsteroidal anti-inflammatory drugs (NSAIDs)
* Use of NSAID or COX-2 within 7 days prior to surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-11; Study Completion 2006-01

PRIMARY OUTCOMES:
Cerebrospinal fluid (CSF) valdecoxib concentration

SECONDARY OUTCOMES:
Plasma valdecoxib concentration
CSF/plasma valdecoxib concentration ratio
CSF and plasma cytokine concentrations
Postoperative opioid consumption
Pain visual analogue scale (VAS) scores

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kharasch, MD PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- University of Washington, Seattle, Washington, United States